CLINICAL TRIAL: NCT06178133
Title: Influencing Factors of the Diagnostic Accuracy of Novel Coronary Functional Evaluation Methods: a Cross-sectional Study
Brief Title: Influencing Factors of the Diagnostic Accuracy of Novel Coronary Functional Evaluation Methods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023683
Record Dates: First submitted 2023-11-14; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FFR: In this single-center cross-sectional study, we included patients with non-acute myocardial infarction who were admitted to the Department of Cardiology at Peking University Third Hospital for FFR testing from January 2019 to December 2021.

SUMMARY:
In this study, patients were retrospectively included, univariate and multivariate analysis of factors affecting their diagnosis inconsistencies was performed, and a new diagnostic model was constructed by logistic regression.

DETAILED DESCRIPTION:
The evaluation of coronary function is becoming more and more important in the guidelines, in which coronary flow reserve (FFR) is the gold standard for diagnosis, but its measurement process requires the application of adenosine, vasodilator, etc. Some patients cannot be measured because of asthma and low blood pressure. A new instantaneous wave-free ratio (iFR), contrastive flow reserve fraction (cFFR) and quantitative flow fraction (QFR) have been developed for the evaluation of coronary function. However, in some patients, the new coronary function evaluation methods were inconsistent with FFR. In this study, patients were retrospectively included, univariate and multivariate analysis of factors affecting their diagnosis inconsistencies was performed, and a new diagnostic model was constructed by logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 80 years old, regardless of gender;
* FFR was detected by coronary angiography;
* The coronary angiography images were clear, meeting the requirements of QFR analysis or detecting iFR, cFFR, and resting pd/pa during the operation.

Exclusion Criteria:

* 1) Coronary artery bypass graft (CABG);
* 2) Atrial fibrillation or flutter;
* 3) Left or right coronary opening lesions;
* 4) Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion criteria and those who did not meet the exclusion criteria were admitted to the Department of Cardiovascular Medicine of Peking University Third Hospital from January 1, 2019 to November 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
the discordance between fractional flow reserve and quantitative flow ratio | When the patient has completed coronary angiography and received a diagnosis
  If FFR≤0.80 and QFR ≤0.8 or FFR > 0.80 and QFR > 0.8 are consistent groups, otherwise they are inconsistent group

CONTACTS AND LOCATIONS:
Overall Officials: Ruitao Zhang, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No